CLINICAL TRIAL: NCT04905017
Title: Early Feasibility Study of the Trisol System
Brief Title: Trisol System EFS Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trisol Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS-10809
Record Dates: First submitted 2021-05-20; First posted 2021-05-27 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-01

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment with the Trisol System (Experimental)
  Interventions: Device: Transcatheter Tricuspid Valve Replacement

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Replacement — Replacement of the tricusupid valve using Trisol System in a transcatheter approach

SUMMARY:
The objective of this early feasibility study is to gain early clinical insight into Trisol system safety and performance to treat patients with moderate or greater tricuspid regurgitation (TR).

DETAILED DESCRIPTION:
A prospective, single-arm, open-label, multi-center early feasibility clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Subject meets the legal minimum age to provide informed consent based on local regulatory requirements.
3. Participant has symptomatic, moderate or greater functional or degenerative tricuspid regurgitation (TR) as determined by the Echocardiography Core Lab assessment of a qualifying transthoracic echocardiogram (TTE) and/or transesophageal echocardiogram (TEE).
4. New York Heart Association (NYHA) Functional Class II to IVa.
5. Participant is deemed at high surgical risk or greater for tricuspid valve surgery and appropriate for transcatheter tricuspid valve replacement as determined by the local Heart Team.
6. Participant adequately treated based upon medical standards, including for coronary artery disease, mitral regurgitation, and Guideline-Directed Medical Therapy (GDMT) for heart failure for at least 30-days prior to index procedure.
7. Male or non-pregnant female.
8. Participant understands the nature of the procedure and provides written informed consent prior to any study specific assessments.
9. Participant is willing and able to comply with the specified study requirements and follow-up evaluations.
10. Participant is anatomically suitable for the Trisol system, including trans-jugular access as per imaging requirements, and is approved by the Subject Screening Committee

Exclusion Criteria:

1. Previous tricuspid valve repair or replacement which may impede proper study device delivery or deployment.
2. Stroke or transient ischemic event within the previous 90 days.
3. Acute myocardial infarction within the previous 90 days.
4. Hemodynamic instability requiring inotropic therapy or mechanical hemodynamic support devices.
5. Untreated clinically significant coronary artery disease requiring revascularization.
6. Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter-defibrillator within the previous 30 days.
7. New or untreated right heart chamber or/and superior vena cava intracardiac mass, thrombus, or vegetation.
8. Systolic pulmonary arterial pressure (sPAP) > 80 mmHg as measured by pulmonary pressure catheter.
9. Severe RV dysfunction with RV Stroke Work Index (RVSWI) g/m2/beat <400 and Pulmonary Artery Pulsatile index (PAPi) <2.
10. Ongoing sepsis, including active endocarditis.
11. Active infection requiring current antibiotic therapy.
12. Known bleeding diathesis or hypercoagulable state.
13. Blood dyscrasias as defined: leukopenia (WBC <3000 cells/mm3), thrombocytopenia (platelet count <50,000 cells/mm3).
14. Active gastrointestinal (GI) bleeding or history of GI bleed within the previous 60 days that would preclude anticoagulation.
15. LVEF <25% as measured by resting echocardiogram within 30 days prior to index procedure.
16. Patients in whom transesophageal echocardiography is contraindicated.
17. Aortic, mitral or pulmonary valve disease (severe stenosis or severe regurgitation) requiring intervention or performed within 90 days prior to enrollment.
18. Severe tricuspid valve stenosis.
19. Need for any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days prior to index procedure.
20. Need for emergent or urgent non cardiac surgery for any reason.
21. Contraindication or known allergy to device components, anticoagulation therapy with a vitamin K antagonist, or to contrast media that cannot be adequately premedicated.
22. History of cardiac transplantation, or participant currently listed for urgent transplant (e.g., UNOS Status 1).
23. Presence of any known life-threatening non-cardiac disease that will limit the subject's life expectancy to less than one year.
24. Contraindication or known hypersensitivity to anticoagulant therapy and/or antiplatelet therapy.
25. Venous anatomy unsuitable for implant delivery.
26. Pacemaker or ICD lead present that would prevent appropriate valve placement.
27. Active COVID-19 infection.
28. Comorbid condition(s) that, in the opinion of the investigator, could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study.
29. Previously enrolled in this study or currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of device-related serious adverse events | Up to 30 days
  Rate of device-related serious adverse events, including death (cardiovascular and non- cardiovascular), MI (MVARC definitions), disabling stroke, life-threatening bleeding (MVARC type III-V), renal failure requiring dialysis, emergency surgery, need for additional surgical procedures due to device failure
Rate of technical success | During procedure
  Technical success: delivery and deployment of the device in the correct position and retrieval of the delivery system.
Rate of procedural success | Up to 30 days
  Procedural success: freedom from emergency surgery or reintervention related to the device or access procedure, without death, stroke, or device dysfunction
Change in TR from baseline | During procedure
  Change in TR from baseline: reduction in TR grade immediately following implantation as compared to baseline TR grade, based on TEE imaging.

SECONDARY OUTCOMES:
Clinical performance endpoints - Change in TR from baseline | At 30 days, 6 months, 12 months
  Change in TR from baseline: reduction in TR grade as compared to baseline TR grade, based on TTE imaging
Clinical performance endpoints - Change in NYHA class | At 30 days, 6 months, 12 months, and then annually
  New York Heart Association (NYHA) functional class: change in NYHA from baseline
Clinical performance endpoints --minute walk test | At 30 days, 6 months and 12 months
  Six-minute walk test: change in distance (m) from baseline
Quality-of-Life: change from baseline as measured by Kansas City Cardiomyopathy Questionnaire | At 30 days, 6 months and 12 months
  Clinical performance endpoints -Quality-of-Life: change from baseline as measured by Kansas City Cardiomyopathy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Isaac George, MD, Principal Investigator — Columbia University
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - Columbia University Medical Center/NYPH, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Main Line Health / Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia Cardiology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No